CLINICAL TRIAL: NCT00415727
Title: Prevention Of Morbidity In Sickle Cell Disease Pilot Phase
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 99NR31
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Sickle Cell Anaemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: auto Continuous Positive Airways Pressure (CPAP) with oxygen supplementation

SUMMARY:
The hypothesis is that in sickle cell anaemia, nocturnal oxyhaemoglobin desaturation, is associated with low processing speed index, and this morbidity can be reduced with overnight auto Continuous Positive Airways Pressure and/or oxygen supplementation.

DETAILED DESCRIPTION:
Intervention: Overnight auto Continuous Positive Airways Pressure (CPAP) with oxygen supplementation if mean overnight oxyhaemoglobin saturation is not >94% after 2 weeks of autoCPAP

ELIGIBILITY:
Inclusion Criteria:

1. Age >4 years.
2. Informed consent with assent in accordance with UK ethical committee(COREC) system must be signed by the patient's parent or legally authorized guardian acknowledging written consent to join the study. When suitable, patients will be requested to give their assent to join the study.
3. Haemoglobin SS (homozygous sickle cell anaemia) diagnosed by standard techniques. Participating institutions must submit documentation of the diagnostic haemoglobin analysis.

Ages: 4 Years to 16 Years | Sex: All
Age Groups: Child
Enrollment: 22
Dates: Start 2006-11

PRIMARY OUTCOMES:
Change in processing speed index

SECONDARY OUTCOMES:
Frequency of pain measured via SMS and pain diary
Adverse events e.g. headache, anorexia, weight loss, nausea, vomiting, reduction in steady state red or white cell count
Change in Blood pressure
Number of omissions on Conners Continuous Performance Test
Change in Chervin sleep Questionnaire
Change in Behaviour Rating Inventory of Executive Function (BRIEF)
Change in number of abnormalities (Adams' criteria) on TCD

CONTACTS AND LOCATIONS:
Overall Officials: Fenella Kirkham, Dr, Principal Investigator — Institute Of Child Health and Great Ormond Street Hospital
Locations (2):
- United Kingdom (2):
  - Neuroscience Unit, Institute of Child Health, London
  - Kings College hospital, London